CLINICAL TRIAL: NCT03913156
Title: Feeding Patterns and Practices in Young Children With PKU During the First Two Years of Life: Acceptability and Efficacy of a New Protein Substitute
Brief Title: Feeding Patterns and Practices in Young Children With PKU During the First Two Years of Life
Acronym: PKU-weaning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B2970
Record Dates: First submitted 2018-08-28; First posted 2019-04-12 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: PKU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Other): Part 1 of the study will recruit subjects who are about to be introduced to a concentrated phe-free protein substitute (i.e. second stage protein substitute) for the first time.
  Interventions: Other: B2970 Metabolic Texture Modified Protein Substitute
- Part 2 (Other): Part 2 of the study will recruit subjects who have already been introduced to a concentrated phe-free protein substitute (i.e. have already transferred from phe-free infant formula onto a second stage protein substitute). This group will be included to evaluate the acceptability of the study product in patients who have already moved onto a second stage protein substitute.
  Interventions: Other: B2970 Metabolic Texture Modified Protein Substitute

INTERVENTIONS:
Other: B2970 Metabolic Texture Modified Protein Substitute — The study product is a powdered phe-free protein substitute supplemented with long chain polyunsaturated fatty acids (LCP's), containing essential and non-essential amino acids, carbohydrate, fat, vitamins, minerals and trace elements and has been designed for use in the management of proven PKU in children aged 6 months to 5 years.
  Other Names: PKU gel

SUMMARY:
In this study the feeding patterns and practices at the introduction of a second stage phe-free protein substitute will be assessed in young children with PKU. This will be compared with the normal weaning process in healthy non-PKU age-matched children. In addition, tolerability and acceptability of the study product will be evaluated in a smaller group of subjects who have already been transferred onto a second stage protein substitute. The study is performed in 3 centers in the United Kingdom.

DETAILED DESCRIPTION:
Part 1:

For subjects with PKU, the study product will be incorporated in the diet as the second stage protein substitute until the subjects are 2 years of age.

The healthy non-PKU age-matched subjects will not have the study product incorporated in their diet in order to be able to compare the weaning experience and nutritional intake of PKU subjects with non-PKU subjects. The healthy subjects will also be part of the study until the subjects are 2 years of age.

Part 2:

All PKU subjects will take the study product for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU identified on screening during the newborn period and requiring a phenylalanine free protein substitute
* Subjects who are about to commence weaning and require a concentrated phe-free protein substitute to meet their total protein requirements and are aged between 4 and 10 months (Part 1)
* Subjects aged under 5 years who have already been fully transferred onto a concentrated phe-free protein substitute and are willing to try the study product for 7 days (Part 2)
* Written informed consent obtained from subject or parents / caregiver
* May or may not have commenced weaning solids (i.e. using normal foods)

Exclusion Criteria:

* Presence of serious concurrent illness
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Any child who has not commenced a second stage protein substitute and is over the age of 10 months
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Any children having taken antibiotics over the previous 2 weeks leading up to the study

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2010-03-15 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Feeding patterns- product intake | up to 2 years
  Actual intake of product and prescribed amount of product [# sachets] will be recorded as documented in diaries.
Feeding patterns - intake other than study product | up to 2 years
  Intakes of standard formulas / breast-milk and normal foods [mL] or [g/day] and [frequency] of breastfeeding, as documented in diaries.
Feeding practices and difficulties by questionnaire; position | up to 2 years
  Feeding practices entered by parents in diaries: the way the child has been fed will be assessed : categories [sitting position e.g on lap, in chair etc]
Feeding practices and difficulties by questionnaire; self feeding | up to 2 years
  Feeding practices entered by parents in diaries; the way the child has been fed will be assessed : [self-feeding; parent feeding]; [type of self feeding: bottle, finger; spoon, fork]
Occurence of Adverse Events [ Safety and tolerability] | up to 2 years
  Occurence of Adverse Events
Gastro-Intestinal symptoms | up to 2 years
  Occurence of GI symptoms [yes/no] for:
  * Mouth Ulcers
  * Tummy upset
  * Harder poos
  * Constipation
  * Softer poos
  * Vomiting
  * Colic
  * Other (free entry)
Product Acceptability yes/no | up to 2 years
  Acceptability questions [yes/no] for:
  * Refuses more than takes
  * Refuses as much as takes
  * Takes more than refuses
  * Spits out product
  * Puts spoon away
  * Holds in mouth but won't swallow
  * Closes mouth on feeding
  * Cries at beginning of feed
  * Cries at end of feed
  * Deliberately spills feed
  * Turns head away
  * Other (free entry)
Blood Phenylalanine control: Phe levels | up to 2 years
  Phe levels [umol/L]
Blood Tyrosine levels | up to 2 years
  Tyrosine levels [umol/L]
Intake of energy and nutritients: Study product | up to 2 years
  Intakes of energy and nutrients from the study product [diet diary; #g product/day]
Intake of energy and nutritients: Weaning | up to 2 years
  Intakes of energy and nutrients from the weaning diet: descriptive information, intakes [g/day]
Intake of energy and nutritients: Weaning | up to 2 years
  Intakes of energy and nutrients from the weaning diet: descriptive information, intakes [# meals or snacks/day]
Anthropometry: weight | up to 2 years
  Weight [g]
Anthropometry: length | up to 2 years
  Length [cm]

SECONDARY OUTCOMES:
Weaning per group (with our without protein substitute) - descriptive | up to 2 years
  Compare the weaning , nutritional intakes [g/day] and metabolic control of infants taking the study product, with historical controls of the same age and weaning stage whose diet did not incorporate a semi-solid second stage protein substitute during the same time period [parent questionnaires]
Anxiety levels of parents - Beck's Anxiety inventory | up to 2 years
  The Beck's Anxiety Inventory, scores on domains [0 not at all - 3 severely]
Coping mechanisms of parents by questionnaire | up to 2 years
  Coping Health Inventory for Parents (scores on domains coping behaviour [3 extremely helpful -0 not helpful]
Parent experience of Feeding via questionnaire | up to 2 years
  Feeding time Parent Questionnaire, experience of parents of their child's feeding time, scores on various domains [0-7]

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Birmingham Children's Hospital
Locations (3):
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, St Luke's Hospital, Bradford
  - JB Russell House, Gartnavel Royal Hospital, Glasgow

REFERENCES:
- See also: Growth, protein, and energy intake in children with PKU taking a weaning protein substitute in the first 2 years of life: a case-control study; Nutrients 2019, 11(3), 552; — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6471165/
- See also: How Does Feeding Development and Progression onto Solid Foods in PKU Compare with Non-PKU Children During Weaning?; Nutrients 2019, 11(3), 529 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6470524/
- See also: Mealtime Anxiety and Coping Behaviour in Parents and Children During Weaning in PKU: A Case-Control Study; Nutrients. 2019 Dec; 11(12): 2857 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6950038/